CLINICAL TRIAL: NCT00377559
Title: Phase II Multicentre Open Label Trial Evaluating the Efficacy and Safety of the Liposomal Doxorubicin (Myocet®) and Docetaxel (Taxotere®) Combination as First-line Treatment of Patients With Metastatic HER2/Neu Negative Breast Cancer
Brief Title: Liposomal Doxorubicin and Docetaxel in HER2 Negative Metastatic Breast Cancer
Acronym: MYOTAX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Cephalon (Industry); Sanofi (Industry)
Responsible Party: Raymond J.P. Schmidt, MD, Stichting (Foundation) BO3
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYOTAX
Record Dates: First submitted 2006-09-15; First posted 2006-09-18 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer; Neoplasm Metastasis
Keywords: Breast cancer; metastatic; cardiotoxicity; liposomal; doxorubicin; docetaxel; HER2/neu negative metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Cardiotoxicity | interventions — Docetaxel; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1. (Experimental): Myocet+docetaxel
  Interventions: Drug: Non pegylated liposomal doxorubicin and docetaxel

INTERVENTIONS:
Drug: Non pegylated liposomal doxorubicin and docetaxel — max. 6 courses
  Other Names: Myocet, Taxotere

SUMMARY:
This is an open phase II multicentre study evaluating the efficacy and safety of the non pegylated liposomal doxorubicin (Myocet®) and docetaxel (Taxotere®) combination as first-line treatment of patients with metastatic HER2/neu negative breast cancer.

DETAILED DESCRIPTION:
Phase II non comparative study, assessing the safety (primarily cardiac safety) and efficacy in patients with locally advanced or metastatic HER2/neu negative breast cancer not yet treated with chemotherapy for metastatic disease.

Myocet and Taxotere will be given for a maximum of 6 cycles. Endpoints: cardiotoxicity (left ventricular ejection fraction decrease and/or symptoms of heart failure), serious other toxicity, disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically documented metastatic or locally advanced metastatic HER2/neu negative breast cancer.
* In the case of previous adjuvant or neoadjuvant chemotherapy with anthracyclines or taxanes, this must have been completed more than 12 months before inclusion.
* In the case of previous adjuvant or neoadjuvant chemotherapy, cumulative anthracycline dose ≤ 360 mg/m2 of doxorubicin or 600 mg/m2 of epirubicin or 75 mg/m2 of mitoxantrone on inclusion.
* Previous endocrine therapy is authorized (endocrine therapy other than goserelin must be stopped before starting treatment).
* Previous radiotherapy is authorized, if discontinued ≥ 4 weeks prior to inclusion in the study and if < 10% of the bone marrow was within the irradiated area.
* Age ≥ 18 years.
* Performance status 0,1, or 2.
* Life expectancy ≥ 3 months.
* Evaluable disease.
* Normal LVEF (multigated acquisition [MUGA] scan or echocardiography).
* Normal haematological, hepatic and renal parameters: neutrophils ≥ 1.5 x 10^9/l; platelets ≥ 100 x 10^9/l; hemoglobin (Hb) ≥ 6 mmol/L; total bilirubin ≤ 1.5 times the upper limit of normal (ULN); transaminases ≤ 2.5 x ULN; alkaline phosphatase ≤ 2.5 x ULN; creatinine ≤ 1.5 x ULN.
* Dated and signed written informed consent.

Exclusion Criteria:

* Previous chemotherapy for metastatic disease.
* History of other cancer, except for cervical carcinoma in situ treated by cone resection or basal cell or squamous cell skin cancer.
* History of congestive heart failure or myocardial infarction ≤ 1 year; cardiac function: NYHA ≥ 2 or LVEF < 50%. Uncontrolled significant heart disease, such as unstable angina.
* Poorly controlled hypertension.
* Performance status 3, 4.
* Symptomatic or progressive brain metastases.
* Active infection or other serious underlying disease.
* Concomitant participation in other clinical trials.
* Pregnant women or nursing mothers; patients of childbearing potential without effective contraception.
* Absolute medical contraindication to the use of corticosteroid premedication.
* Allergy to polysorbate 80, doxorubicin, or egg lecithin.
* NCI-CTC grade > 1 peripheral neuropathy.
* Patients not able to comply with regular medical follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-05; Primary Completion 2009-11 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Cardiotoxicity (definite or probable cardiac death) | treatment period
Signs or symptoms of congestive heart failure (CHF), New York Heart Association (NYHA) class III-IV | treatment period
Decline in left ventricular ejection fraction (LVEF) of ≥ 5% to < 50% with mild signs or symptoms of CHF (NYHA class < III) | treatment period
Decline in LVEF of ≥ 10% to < 50% without signs or symptoms of CHF | treatment period

SECONDARY OUTCOMES:
Frequency and severity of intercurrent events according to the National Cancer Institute - Common Terminology Criteria (NCI-CTC) classification | treatment period
Response rate | treatment period
Median time to progression | treatment period
Progression free survival | treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Laurence J. van Warmerdam, MD, PhD, Principal Investigator — Catharina Ziekenhuis
Locations (10):
- Netherlands (10):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Wilhelmina Ziekenhuis, Assen
  - Catharina-Ziekenhuis, Eindhoven
  - Ziekenhuis Walcheren, Flushing
  - Ikazia Ziekenhuis, Rotterdam
  - Sint Elisabeth Ziekenhuis, Tilburg
  - Mesos Medisch Centrum, Utrecht
  - Maxima Medisch Centrum, Veldhoven
  - VieCuri MC, Venlo
  - Streekziekenhuis Koningin Beatrix, Winterswijk